CLINICAL TRIAL: NCT06697912
Title: Observational Study of Breathing and Flows in Bubble-CPAP Used With the RAM Cannula Interface in Newborn Infants
Brief Title: Airway Flow of RAM Cannula With BCPAP in Infants
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Thomas Drevhammar, Ass. Prof. (Docent), Karolinska Institutet
Other Study IDs: 1758 CN/PS
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Distress Syndrome, Newborn; Infant, Premature, Diseases; Infant, Newborn, Diseases
Keywords: Continuous Positive Airway Pressure; Respiratory Therapy
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Infant, Premature, Diseases; Infant, Newborn, Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infant treated with bubble CPAP and receiving blended air/oxygen

SUMMARY:
The RAM Cannula interface is used as routine interface for newborn infants receiving CPAP treatment for respiratory distress. Compared to the standard systems that have been used for more than 50 years, the interface has high resistance and has not been extensively studied. The delivered quality of the CPAP support is likely to be negatively affected by the interface resistance.

We hypothesise that exhalations through the device is uncommon and that the interface resistance restricts flow from the patient. If expiratory flows are uncommon the RAM interface provide support clinically comparable to other systems based on unidirectional flow such as humidified high-flow cannula.

This is a cross-sectional, observational study (no intervention) in newborn infants that are clinically stable and on respiratory support with the RAM interface connected to a bCPAP circuit. This is the most common support in the Phu San neonatal unit. The time needed for data collection is short and collection is expected to take approximately five minutes (less than 15 minutes) in a quiet infant. The collection can be planned to minimize disturbances for the infant, parents and staff. For example, the busiest times of the day can be avoided to not intervene with daily care, ward rounds or examinations of the infant.

Data on flow and pressure will be collected within the respiratory support circuit at the connection to the RAM interface. The measurements are passive, and no tests or manipulation of the infant is planned. There will be brief interruptions (<1 min) in respiratory support when the meters are connected. Similar interruptions are very common and occurs several times per day during normal care.

Data will be collected in case report forms (CRF) with REDCap electronic data capture tool. All personal identifiers will be removed before data export from REDCap and further analysis only using enrolment numbers.

Background variables describing the pregnancy, delivery and the infant will be collected. We also will record details of the RAM-cannula interface, such as size, protective dressing, gastric feeding tube, obvious leak at nares and mouth.

During the measurement the infant will be monitored for vital signs and any problems will be addressed and recorded. This includes oxygen need, CPAP support and breathing problems. The flow and pressure data for one minute of quiet breathing will be stored locally with the enrolment number as identifier. The analysis after collection of flow and pressure will include average flow in the CPAP circuit, the flow to the patient, average absolute leak and delivered pressure. If a variation with breathing can be seen this will be described. These output variables directly relate to the research questions.

1. What flows and pressure can be observed in the breathing circuit? [Measured average flows, pressure and variability between patients]
2. Do infants exhale through the RAM interface? [Measured expiratory flows at the interface]
3. What is the level of leak for the interface? [Measured absolute leak]

The RAM cannula interface has been widely introduced but is not CE-marked for CPAP support. It has an advantage of being more comfortable and light weight with less nasal injury in most trials. The high resistance of the RAM interface has been discussed as problematic by several authors, but the clinical importance is not known. Comparing RAM interface to other CPAP interfaces in clinical trials is difficult and, if RAM has a treatment effect similar to HHFNC, very large trials of high quality would be needed.

The described study will generate new knowledge on the RAM interface by describing patient flow through the interface and illustrate the importance of resistance and leak. The study is not strictly a physiological study but investigate flow in an airway interface. The most likely outcome is that exhalation is uncommon, and this would support that the RAM interface has more similarities with HHFNC than conventional CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Phu San Hanoi Hospital Neonatology Unit
* Support with bubble CPAP and RAM interface
* Quiet and stable spontaneous breathing
* Investigation team available

Exclusion Criteria:

* Problems with routine CPAP care
* Major congenital malformation
* Known syndrome or neuromuscular disease
* Circulatory instability with inotropes
* Oxygen need >50% or CPAP >10 cm H2O
* Surfactant given the last 6 hours or expected to be needed the next 6 hours
* Expected to need NIPPV or intubation within 6 hours
* Recently extubated (<24 h)
* Recent large surgical procedure (<5 days)
* Nasal wound or irritation that hurts or is at risk of worsening during study

Ages: 0 Hours to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants treated with RAM interface and bubble CPAP system that are clinically stable, spontaneous breathing and not expected to need any urgent interventions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Airway flow in RAM interface | 60 seconds
  Average airway flow (L/min) in a quiet breathing infant

SECONDARY OUTCOMES:
Pressure at Y-piece connector of RAM interface | 60 seconds
  Average pressure (cm H2O) over 60 seconds in a quiet breathing infant
Fresh gas flow to Y-piece connector for RAM interface | 60 seconds
  Average flow (L/min) over 60 seconds in a quiet breathing infant
Exhalation through Y-piece connector for RAM interface | 60 seconds
  Number of breaths (ratio) with an expiratory flow of (duration >0.1 ms) over 60 seconds in a quiet breathing infant

OTHER OUTCOMES:
Adverse events | 1 hour
  Any adverse events during the measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Phu San Hanoi Hospital, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study will be available from the principal investigator on reasonable request after publication of results.